CLINICAL TRIAL: NCT01880749
Title: Exploring the Activity of RAD001 in Vestibular Schwannomas and Meningiomas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12-02808
Record Dates: First submitted 2013-06-11; First posted 2013-06-19 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Neurofibromatosis Type 2; Vestibular Schwannomas; Meningiomas
MeSH Terms: conditions — Neurofibromatosis 2; Neuroma, Acoustic; Meningioma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RAD001 (Experimental): RAD001 taken by mouth 10mg daily for 10 days before surgery
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001
  Other Names: Everolimus

SUMMARY:
The primary objective is to estimate the proportions of vestibular schwannomas (VS) and meningiomas after 10 days of exposure to the study drug RAD001 at a dose of 10 mg daily, as determined by immunohistochemistry. This is a "phase 0" PK (pharmacokinetic) and PD (pharmacodynamic) study of RAD001 in patients with Neurofibromatosis Type 2-related and sporadic VS and meningiomas. Enrolled patients will take RAD001 prior to a scheduled VS or meningioma surgery, and blood and tissue samples will be obtained for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must satisfy all of the following eligibility criteria:
* Karnofsky performance status (KPS) ≥ 60%
* Absolute neutrophil count ≥ 1,000/mm³ (unsupported)
* Platelet count ≥ 100,000/mm³ (unsupported)
* Hemoglobin ≥ 8 g/dl (transfusion support allowed)
* Creatinine ≤ 1.5 times upper limit of normal (ULN*) OR corrected glomerular filtration rate ≥ 70 ml/min
* Total bilirubin ≤ 1.5 times ULN*
* ALT ≤ 2.5 times ULN*
* Serum albumin ≥ 2 g/dl
* INR < 1.3 (or < 3 on anticoagulants)
* Patients taking a cholesterol-lowering agent must be on a single medication and on a stable dose for at least 4 weeks
* Fasting serum cholesterol ≤ 300 mg/dl OR ≤ 7.75 mmol/l AND fasting triglycerides ≤ 2.5 times ULN*.
* Fully recovered from acute toxic effects of any prior chemotherapy, biological modifiers or radiotherapy
* Any neurologic deficits must be stable for ≥ 1 week
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test. The anti-proliferative activity of this experimental drug may be harmful to the developing fetus.
* Able to provide written informed consent

Exclusion Criteria:

* Patients with any of the following are ineligible for this research study:
* Patients with VS or meningiomas deemed very high surgical risk for stroke and/or other complications by the attending surgeon, such as meningiomas with major vascular or dural sinus infiltration.
* Patients with serious concurrent infection or medical illness, which would jeopardize the ability of the patient to receive the treatment outlined in this protocol with reasonable safety.
* Symptomatic congestive heart failure or unstable angina pectoris.
* Uncontrolled diabetes, as defined by fasting serum glucose >1.5 times ULN*.
* Current active hepatic or biliary disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis (with exception of patients with Gilbert's syndrome and asymptomatic gallstones).
* History of hepatitis B or C. Note: A detailed assessment of hepatitis B/C medical history and risk factors must be done at screening for all patients. HBV serology, DNA and/or HCV RNA PCR testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection. If no positive medical history for risk factors, serology is not required.
* Seropositivity or DNA/RNA positivity for hepatitis B or C, with the exception of patients who have received prior Hepatitis B vaccination and are Anti-HBs positive only.
* Known HIV seropositivity
* Neurologic deficits that are rapidly progressing: all neurologic signs and symptoms must have been stable for a week prior to first dose
* Patients who are pregnant or breast-feeding. The anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant.
* Anti-tumor therapy (i.e. chemotherapeutics or investigational agents or immunotherapy) within 4 weeks prior to enrollment
* Radiation therapy to a study target lesion within 6 months
* Prior therapy with mTOR inhibitors, including sirolimus, temsirolimus, deforolimus within 6 months prior to enrollment
* Known hypersensitivity to RAD001 or other rapamycins (sirolimus, temsirolimus, deforolimus)
* Patients with a concurrent malignancy
* Patients treatment with systemic steroids or another immunosuppressive agent. Patients with endocrine deficiencies are allowed to receive physiologic or stress doses of steroids if necessary.
* Patients cannot receive CYP3A4 inhibiting drugs including antibiotics (clarithromycin, erythromycin, troleandomycin), anti-HIV agents (delaviridine, nelfinavir, amprenavir, ritonavir, indinavir, saquinavir, lopinavir), antifungals (itraconazole, ketoconazole, fluconazole at doses > 200 mg/day, voriconazole), antidepressants (nefazodone, fluovoxamine), calcium channel blockers (verapamil, diltiazem) oramiodarone
* Patients should avoid CYP3A4 inhibiting foods including grapefruit and Seville orange juice.
* Patients cannot receive CYP3A4 inducing anticonvulsants including carbamazepine, felbamate, phenobarbital, phenytoin, primidone and oxcarbazepine, or other CYP3A4 inducers such as St. John's Wort
* Patients who previously received CYP3A4 inducers or inhibitors must have discontinued these medications within at least 1 week prior to study entry and can re-start them 1 week post-operatively (or earlier if determined to be of clinical benefit, as determined by the treating physician).

  * of institutional norms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Proportions of VS and meningiomas after exposure to RAD001 | 10 days
  1) To estimate the proportions of VS and meningiomas with complete inhibition of phospho-S6 after10 days of exposure to RAD001 at a dose of 10 mg daily, as determined by immunohistochemistry. This endpoint was chosen based on prior pharmacodynamic data from a published trial, showing complete inhibition of phospho-S6 in solid tumor tissue of patients treated with RAD001 and our own preliminary data confirming baseline phospho-S6 expression in VS and meningiomas.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Nicolaides, MD, Study Chair — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States